CLINICAL TRIAL: NCT01948479
Title: Prevention of Foot Ulcer Recurrence in People With Diabetes Using an In-shoe Pressure Measurement Technology: A Randomised Control Trial Feasibility Study
Brief Title: Insole Optimisation for Ulcer Prevention: a Feasibility Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Plymouth (Other)
Collaborators: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Joanne Paton, NIHR Clinical Research Fellow, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PatonRCT02
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Diabetic; Neuropathic; Past Ulceration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insole optimised with inshoe analysis (Experimental)
  Interventions: Device: Optimised instant offloading insole
- Routine insole provision (Active Comparator)
  Interventions: Device: Optimised instant offloading insole

INTERVENTIONS:
Device: Optimised instant offloading insole

SUMMARY:
Insoles are designed to reduce increased loads and re-ulceration risk in patients with diabetes. The investigators previous research findings suggest that an instant insole solution may benefit some, but effectiveness is difficult to predict. The investigators propose a feasibility study using in-shoe pressure analysis to optimise the protective effect of insoles and footwear with the aim of reducing re-ulceration rates.

Early indications from exploratory case studies within the real world clinical setting suggest that by implementing the investigators previous published research findings the investigators can optimise effectiveness and reduce outcome variability of protective footwear and insoles provided to patients at risk of re-ulceration.

However a further randomised control trial is necessary to evaluate the effectiveness of in-shoe pressure analysis in reducing re-ulceration rates within the NHS setting. The proposed feasibility study will recruit 20 participants from the multidisaplinary diabetic foot clinic Derriford Hospital and allocate them to either 1) Routine insoles and footwear provision or 2) Routine insole and footwear provision, and temporary insole provision with optimisation. The findings from the feasibility study will inform protocol development for a larger clinical trial. The results of the feasibility study will be used to strengthen a protocol for a grant application to conduct the main RCT. A secondary output from the pilot study will be the dissemination of findings in a peer reviewed journal and at conference.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 30 years or above
* Diagnosed with Diabetes Mellitus
* Recently healed/healing target ulcer on the weight-bearing surface of the foot
* Neuropathic (Mild to moderate DPN defined as insensitivity of a 10 g monofilament at 1-3 sites in the following locations: hallux, 1st, 3rd, and 5th metatarsal heads (Boulton AJ, Armstrong DG, Albert SF, Frykberg RG, Hellman R, Kirkman MS, Lavery LA, Lemaster JW, Mills JL Sr, Mueller MJ, Sheehan P, Wukich DK: Comprehensive foot examination and risk assessment: a report of the task force of the foot care interest group of the American Diabetes Association, with endorsement by the American Association of Clinical Endocrinologists. Diabetes Care 2008;31:1679-1685)
* Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply: Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* None healing foot ulcer at another site that requires targeted off-loading.
* Unable to walk 5 metres with/without walking aid
* Peripheral vascular disease (non-re-constructible vascular disease as determined by arterial duplex and clinically assessed by a vascular consultant)
* Unwilling to wear therapeutic footwear
* Where amputation has been part of the current episode of care and includes ulceration site.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
ulcer recurrence rates | 6 months

SECONDARY OUTCOMES:
peak pressure reduction with the addition of the intervention | Issue and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Derriford Hospital, Plymouth, Devon, United Kingdom